CLINICAL TRIAL: NCT05200884
Title: A Comparison the Effectiveness of Anesthesia With Lidocaine 2% or Articaine 4% in Children With Molar Incisor Hypomineralisation (MIH)
Brief Title: Local Anesthesia With Lidocaine or Articaine for Molars Affected by MIH
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tishreen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Tishreen U _pediatricDentistry
Record Dates: First submitted 2021-12-15; First posted 2022-01-21 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-01

CONDITIONS: Molar Incisor Hypomineralisation
Keywords: the local anesthesia; Lidocaine 2%; Articaine 4%; children; MIH molars.
MeSH Terms: conditions — Molar Hypomineralization

STUDY DESIGN:
Intervention Model Description: A randomized, controlled, crossover, double-blind clinical study, Comparison of articaine 4% and lidocaine 2%
Who Masked: Participant, Investigator
Masking Description: The participant will be blinded, the drug administrator will be blinded too, and the investigator who will give the treatment and explain the pain scale to the participant and ask him\her to point to the face that fits the degree of his pain that associated with the drug administration will also be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- : A (Lidocaine 2%) (Active Comparator): 20 children will be injected with 1 ml of lidocaine 2% with epinephrine. each one received lidocaine2% at his\her ﬁrst or second visit.
  Half of the total number of injections for 20 children i.e. 20 injections will be distributed randomly to the two drugs using the randomization table
  Interventions: Drug: Lidocaine 2%
- B (Articaine 4%) (Experimental): 20 children will be injected with 1 ml of Articaine 4% with epinephrine. each one received articaine 4% at his\her ﬁrst or second visit.
  Half of the total number of injections for 20 children i.e.20 injections will be distributed randomly to the two drugs using the randomization table
  Interventions: Drug: Articaine 4%

INTERVENTIONS:
Drug: Lidocaine 2% — The child will be injected with lidocaine 2% and After 10 minutes the treatment will be completed , Pain during injection and treatment will be assessed using the FLACC scale and pain after injection and treatment will be evaluated using the Wong-Baker FACES pain rating scale
  Other Names: A
  Arms: : A (Lidocaine 2%)
Drug: Articaine 4% — The child will be injected with 4% Articaine and After 10 minutes the treatment will be completed , Pain during injection and treatment will be assessed using the FLACC scale and face scale
  Other Names: B
  Arms: B (Articaine 4%)

SUMMARY:
Aims: Comparison of injection pain with lidocaine and articaine in children with MIH .

Comparison of the efficacy of lidocaine and articaine during treatment of MIH molars.

Design: A randomized, controlled, crossover, double-blind clinical study including twenty cooperative children, aged 6-12years old

DETAILED DESCRIPTION:
Background and Aims: Effectively achieving anesthesia is one of the difficulties a dentist faces when treating MIH molar There are no studies comparing the effectiveness of lidocaine and articaine in MIH molar Design: A randomized, controlled, crossover, double-blind clinical study including twenty cooperative children , aged 6-12 years old Each child will receive either lidocaine or articaine at their ﬁrst or second visit.

ELIGIBILITY:
Inclusion Criteria:

* Absolute positive or positive behavior according to the Frankel Scale.
* Healthy, both physically and mentally.
* Do not take medications that interfere with the assessment of pain within 24 hours prior to treatment.
* A child with a MIH-affected mandibular permanent first molar on the right and left sides .

Exclusion Criteria:

* Teeth with non-response pulpitis Inflammation at the injection site.
* Allergy to the substances used in anesthesia.
* Presence of general or developmental medical conditions.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2022-01-22 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
dental pain | during the injection of local anesthesia
  evaluated by outcome assessor using the Faces, Legs, Activity, Cry, Consolability Behavioral Pain Rating Scale ( FLACC scale ) ( a behavioral pain assessment scale which has five criteria face, legs, activity, cry, consolability ,which are each assigned a score of 0, 1 or 2.Total score of scale is summed in range 0 to 10, where: 0=relaxed and comfortable; 1-3=mild discomfort; 4-6=moderate pain; 7-10=severe pain)..
dental pain | Immediately after the injection of local anesthesia
  self assessment pain by the children using Wong-Baker faces pain rating scale (a scale shows a series of faces ranging from a happy face at 0, or "no hurt", to a crying face at 10,which represents "hurts like the worst pain imaginable" )
dental pain | during treatment
  evaluated by outcome assessor using the Faces, Legs, Activity, Cry, Consolability Behavioral Pain Rating Scale ( FLACC scale ) ( a behavioral pain assessment scale which has five criteria face, legs, activity, cry, consolability ,which are each assigned a score of 0, 1 or 2.Total score of scale is summed in range 0 to 10, where: 0=relaxed and comfortable; 1-3=mild discomfort; 4-6=moderate pain; 7-10=severe pain)..
dental pain | Immediately after the treatment
  self assessment pain by the children using Wong-Baker faces pain rating scale (a scale shows a series of faces ranging from a happy face at 0, or "no hurt", to a crying face at 10,which represents "hurts like the worst pain imaginable" )

CONTACTS AND LOCATIONS:
Overall Officials: Nabih Raslan, Dr, Study Chair — Tishreen University; Mai Haidar, Dr, Principal Investigator — Tishreen University
Locations (1):
- Tishreen University, Latakia, Syria

IPD SHARING:
Plan to Share IPD: Undecided
up to date, there is no decision about IPD sharing.

REFERENCES:
- [Derived] Haidar M, Raslan N. Comparative study of articaine 4% versus lidocaine 2% in the local anesthesia of permanent mandibular first molars affected by MIH: a randomized controlled trial. Eur Arch Paediatr Dent. 2023 Oct;24(5):621-630. doi: 10.1007/s40368-023-00827-w. Epub 2023 Aug 1. PMID 37526883